CLINICAL TRIAL: NCT02180113
Title: Feasibility and Performances of Spleen Stiffness Measurement as Surrogate Marker for Oesophageal Varices in Cirrhotic Patients.
Brief Title: Spleen Stiffness Measurement With FibroScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M116
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Cirrhosis
Keywords: Cirrhotic patients; Fibroscan; Liver Stiffness Measurement; Oesophageal Varices; Portal Hypertension; Spleen Stiffness Measurement
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan® (Other): Fibroscan® is an active non implantable medical device using ultrasound. It has been designed to measure liver stiffness in a painless, rapid and non invasive manner. It is a diagnostic aid tool. In this study, Spleen Stiffness Measurement will be assessed using a dedicated FibroScan® device which has been developed specifically to assess spleen stiffness.
  Interventions: Device: Fibroscan® examination

INTERVENTIONS:
Device: Fibroscan® examination — Each patient undergo 1 LSM and at least 1 SSM (2 in more if the patient accept to participate at the ancillary study (intra and inter operator reproducibility of SSM).

SUMMARY:
FibroScan® (Echosens, Paris, France) is an active non implantable medical device marketed in Europe since December 2003 and is currently used in many countries. FibroScan® is an ultrasound-based vibration-controlled transient elastography (VCTE™) device dedicated to liver stiffness measurement (LSM).

Several clinical studies have shown the accuracy of LSM by FibroScan® to predict liver fibrosis.

Some other studies have already shown the good correlation between LSM, assessed by FibroScan® based on VCTE™ technology, and the presence of portal hypertension (PHT).

PHT is a clinical condition characterized by a high blood pressure in the portal vein and its tributaries and it is defined as a gradient between portal and systemic blood pressure > 6 mmHg.

The development of oesophageal varices (OV) in cirrhotic patients, as well as their potential bleeding, represent one of the most severe and life-threatening complication of cirrhosis.

Upper endoscopy is the best diagnostic tool for detecting the presence of OV, gastric varices or congestive gastropathy, for estimating the grade of OV and for the recognition of the presence of red color signs and wale marks or other indicators of high risk for bleeding.

However these two methods are quite invasive and associated with some risks; at the same time, not all cirrhotic patients present OV at endoscopic screening.

The aim of this study is the validation of SSM, assessed by a FibroScan® with acquisition parameters and algorithm optimized for SSM, as surrogate noninvasive marker for the presence of OV in liver cirrhosis patients.

ELIGIBILITY:
Inclusion Criteria:

* All groups

  * Both gender, 18-79 years old
  * Patient able to give written informed consent form
  * Patient affiliated to a social security system.
* Case group

  * Patient with chronic liver disease due to: hepatitis C virus, hepatitis B virus or Alcoholic Liver Disease and liver stiffness ≥ 14 kPa
  * Patient with the following examination within 3 months of LSM and SSM: ultrasound examination, blood examination, gastroscopy examination and eventually an hepatic venous pressure gradient examination
* Control groups

  * Patient with chronic liver disease due to: HCV, HBV or Alcoholic Liver Disease and liver stiffness < 14 kPa
  * Patients without chronic liver disease (Healthy Control subgroup)

Exclusion Criteria:

* Patient unable or unwilling to provide written informed consent.
* Consuming illness (HIV infection, malignancy).
* Associated comorbidities: NASH, hemochromatosis, primary sclerosing cholangitis, primary biliary cirrhosis.
* Antiviral treatment during the two months before inclusion.
* Pacemaker or heart defibrillator.
* Pregnancy.
* Liver transplantation.
* BMI>35 kg/m2.
* Serum Transaminases > 250 IU/L.
* History of / or current βblockers treatment of OV.
* Presence of ascites.
* Previous endoscopic treatment of OV.
* Patient with acute alcoholic hepatitis and associated jaundice (generally defined by total bilirubin ≥ 50 µmol/l).
* Patient with hepatocellular carcinoma (HCC).
* Unable or unwilling to undergo a liver stiffness measurement, a spleen stiffness measurement, an ultrasound examination, a blood examination or a gastroscopy examination.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2012-03; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Selection of patient with cirrhosis using LSM ≥ 14 kPa (kilopascal) | Up to 36 month

SECONDARY OUTCOMES:
Diagnosis of large OV with an sensitivity of 95% and an acceptable lower bound of 85% | Up to 36 month

OTHER OUTCOMES:
Prevalence of patients with large OV in cirrhotic patients: 30% | Up to 36 month

CONTACTS AND LOCATIONS:
Overall Officials: Davide FESTI, Pr., Principal Investigator — Department of Clinical Medicine, Policlinico S. Orsola Malpighi, Bologna, Italy; Horia STEFANESCU, Dr., Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy, Clu-Napoca, Romania; Victor de LEDINGHEN, Pr., Principal Investigator — Hôpital Haut-Lévêque, Service Hépato-gastroentérologie et Oncologie digestive, Pessac, France; Paul CALES, Pr., Principal Investigator — CHU, Service Hépato-gastroentérologie, Angers, France; Mirella FRAQUELLI, Dr., Principal Investigator — Seconda Divisione di Gastroenterologia Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milano, Italy; Nathalie CARRIE-GANNE, Pr., Principal Investigator — Hôpital Jean Verdier, Service Hépato-gastroentérologie, Bondy, France
Locations (7):
- France (3):
  - CHU, Service Hépato-gastroentérologie, Angers
  - Hôpital Jean Verdier, Service Hépato-gastroentérologie, Bondy
  - Hôpital Haut-Lévêque, Service Hépato-gastroentérologie et Oncologie digestive, Pessac
- Italy (2):
  - Department of Clinical Medicine, Policlinico S. Orsola Malpighi, Bologna
  - Seconda Divisione di Gastroenterologia Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico,, Milan
- Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Romania
- Royal Free Hospital, Pond Street, London, United Kingdom

REFERENCES:
- [Derived] Stefanescu H, Marasco G, Cales P, Fraquelli M, Rosselli M, Ganne-Carrie N, de Ledinghen V, Ravaioli F, Colecchia A, Rusu C, Andreone P, Mazzella G, Festi D. A novel spleen-dedicated stiffness measurement by FibroScan(R) improves the screening of high-risk oesophageal varices. Liver Int. 2020 Jan;40(1):175-185. doi: 10.1111/liv.14228. Epub 2019 Sep 11. PMID 31444849